CLINICAL TRIAL: NCT06532175
Title: Effects of Su Jok Seed Therapy Application on Pain, Anxiety and Psychological Resilience in Patients Hospitalized in the Oncology Ward
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MusAlparlan U
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Cancer Pain
Keywords: su-jok; cancer patients; anxiety; pain; Psychological resilience
MeSH Terms: conditions — Neoplasms; Cancer Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Su-jok Therapy Group /EXPERIMENTAL GROUP (Experimental): Providing a comfortable position considering the individual's limitations. In order for the hands not to be cold, the researcher will warm them by rubbing them together and will plan to grasp the patient's hand.
  The individuals' pain areas will be determined and reflection points corresponding to these areas on the yin and yang sides will be determined.
  The individual will be asked to state when they experience pain and pulling sensations at the points touched by the applicator.
  Determining painful reflection points on the back of the individual's hand When each reflection point is determined, green mung bean will be placed on the relevant point and fixed with a plaster band. The same procedure will be applied to all painful points until the individual states that there are no more painful points The point where the seed is fixed will be massaged for 30 minutes. The individual will be helped to take a comfortable position.
  Interventions: Device: Su-Jok
- Control Group (No Intervention): No intervention will be made. Data will only be collected when the participant participates in the study, one month after participating in the study, and 2 months after participating in the study.

INTERVENTIONS:
Device: Su-Jok — Su-jok seed therapy
  Other Names: Su-jok seed therapy
  Arms: Su-jok Therapy Group /EXPERIMENTAL GROUP

SUMMARY:
The aim of this clinical trial is to determine the effects of su jok seed therapy on pain, anxiety and psychological resilience in patients hospitalized in the oncology ward. This study seeks answers to the following questions; Does su jok seed therapy affect the pain levels of cancer patients? Does su jok seed therapy affect the anxiety levels of cancer patients? Does su jok seed therapy affect the Psychological resilience levels of cancer patients? There will be an experimental and control group in the study and the effectiveness of sujok application will be examined.

A total of 8 sessions of su jok seed therapy will be applied to the experimental group, twice a week for a month. No intervention will be made to the control group.

Individuals over 18 years old, without communication problems and diagnosed with cancer will be included in the sample.

DETAILED DESCRIPTION:
Location of the study:

Research data will be collected in the oncology unit of Muş State Hospital.

Time of the study:

Research data will be collected between June 15 and December 31, 2024.

Research universe, sample, research group:

The research universe will consist of patients who apply to the oncology service in the hospital where the study is conducted and receive treatment. Before determining the sample of the study, a priori power analysis was performed in the GPOWER 3.1.9.7 Package Program based on the "Dependent Groups t Test". It was determined that the number of samples required for the study to exceed 80% with a 95% confidence interval, a significance level of 0.05, and a medium effect size, was 68 people, with 34 people in each group. In order for the study to exceed 80% power and considering possible data losses, the total sample number was determined as N: 80, with 40 in the intervention group and 40 in the control group.

Required manpower for the research:

Güzel Nur Yıldız: Analysis, findings and writing the method Arzu KARAKAYA: Data collection (she received the Su Jok certificate by attending the Su Jok certification training given by the International Su Jok Association), discussion writing, introduction writing and general organization.

Research method and data collection tools:

"Descriptive Characteristics Form" and "State Anxiety Scale", "Brief Psychological Resilience Scale" and "Visual Comparison Scale" will be used as data collection tools.

Descriptive Characteristics Form This form, prepared by the researcher based on literature, includes questions such as the age, gender, socioeconomic level and educational status of the patients.

State Anxiety Scale: The State Anxiety Inventory expresses how the participant feels at a certain moment and period. According to the severity of the emotions and behaviors expressed in the items of the scale, one of the options '(1) None, (2) A Little, (3) A Lot, (4) Completely' is selected (Karadağ & Uğur, 2021).

Brief Psychological Resilience Scale (BRS: The Brief Psychological Resilience Scale (BRS) is a 5-point Likert-type measurement tool consisting of six items developed to measure the psychological resilience of individuals. The scale was adapted to Turkish by Doğan in 2015. When the scale is graded, items 2, 4 and 6 are scored reversely. A high score from the scale indicates a high level of psychological resilience, while a low score indicates a low level of psychological resilience (Doğan 2015). A score between 6-11 indicates a low level, 12-22 indicates a medium level and 23-30 indicates a high level. The Cronbach Alpha coefficient calculated in the validity and reliability study of the scale is 0.79 (Doğan, 2015) Visual Analog Scale (VAS): Developed by Freyd in 1983, the scale is a reliable measurement tool developed to measure the pain levels of individuals. The scale is simple, attractive, can be filled out quickly and can be scored easily (Freyd, 1923). There are subjective descriptive statements at both ends of a 10-cm ruler.

RANDOMIZATION Patients applying to the oncology unit will be separated into single and double according to the order of application. Single patients will form the experimental group, and double patients will form the control group. An application for a Clinical Trials ID number will be made after the ethics committee is received.

Control group: No intervention will be made to this group. When the participants participate in the study, after one and two months, they will be asked to fill out the "State Anxiety Scale", "Brief Resilience Scale" and "Visual Comparison Scale".

Experimental group: This group will be given su jok therapy using green mung bean seeds. A total of 8 sessions (twice a week for 4 weeks) of therapy will be applied. Green mung bean seeds will be placed on a certain point of the patient's hand and taped. After two hours, they will be asked to remove and throw it away. When the participants participate in the study, after one and two months, they will be asked to fill out the "State Anxiety Scale", "Brief Resilience Scale" and "Visual Comparison Scale".

In the last stage, the data obtained will be compared within and between groups.

Su Jok Application Process Steps The researcher received the Su Jok certificate by attending the Su Jok certification training given by the International Su Jok Association. Green mung bean seeds were used in the research. The seed will be purchased from an institution that is certified as organic and has an entrepreneurial certificate. Su Jok will be applied to the reflection points on the hand based on the painful area of the individual. The painful areas will be determined with the applicator and green mung bean will be placed in these areas. It is planned to apply a circular massage to the areas where the seeds are located for 30 minutes and to carry out all the steps as follows.

Before the Procedure • Informing the individual about the procedure.

Providing hand hygiene.

A comfortable position will be provided considering the individual's limitations.

In order for the hands not to be cold, the researcher will warm them by rubbing them together and the patient's hand will be grasped.

Su Jok applicator has been taken. Procedure Order: Individuals' pain areas will be determined and reflection points corresponding to these areas on the yin and yang sides will be determined.

The individual will be asked to state when they experience pain and pulling sensations at the points touched by the applicator.

Determining painful reflection points on the back of the individual's hand

* When each reflection point is determined, green mung bean will be placed on the relevant point and fixed with a plaster band. The same procedure will be applied to all painful points until the individual states that there are no more painful points
* Massage will be applied to the point where the seed is fixed for 30 minutes. After the Procedure • The individual will be helped to take a comfortable position.

Hands will be washed.

Data Collection:

Research data will be collected by the researcher using the face-to-face interview method. First, individuals who will participate in the study will be determined and individuals will be randomly divided into experimental and control groups. Participants in the experimental and control groups will first fill out the "Voluntary Consent Form", "State Anxiety Scale", "Brief Resilience Scale" and "Visual Comparison Scale". The experimental group will receive su jok therapy with green mung bean twice a week for a total of 4 weeks (8 sessions in total). The control group will not receive any intervention. Participants will fill out the "State Anxiety Scale", "Brief Resilience Scale" and "Visual Comparison Scale" again after one month and two months. The researchers will not perform any invasive procedures. Su jok therapy with fresh yeast seed is performed by placing seeds on certain points on the hands of individuals. Individuals will not swallow this seed, they will just put it in a certain place on their hand, tape it and wait for two hours, then take it out and throw it away. Therefore, no invasive procedure will be performed on individuals in this therapy. In order to collect the data, written permission will first be obtained from the institutions where the research is conducted. Before the interview with the individuals, explanations will be made about the purpose and objectives of the research, the benefits to be obtained from the research, and the time they will spend for the interview, and their verbal consent will be obtained. In the Google Forms method, an explanation will be made on the first page of the form and consent will be obtained. The data will be collected in an average of 15-30 minutes.

Data analysis:

The data will be evaluated in the SPSS (Statistical Package for Social Sciences for Windows, Version 22.0) package program. In the evaluation of the data, the statistical significance value will be accepted as 0.05, the Type 1 error will be kept as 5%, and the evaluation will be made with a 95% confidence interval. Skewness and Kurtosis values will be examined in order to determine whether the measurements show a normal distribution. According to Skewness, the range of +1 -1 is normal, and the range of +2 -1 is normal for Kurtosis. Data will be analyzed in light of this information. In intergroup comparisons, the t-test will be used for independent groups in measurements showing normal distribution, and the Mann Whitney U test will be used for measurements not showing normal distribution. In intragroup pretest posttest score comparisons, the t-test will be used for dependent samples in measurements showing normal distribution, and the Wilcoxon test will be used for measurements not showing normal distribution. In order to determine the difference in repeated measurements, the single factor anova will be used for Renewed Measurements in measurements showing normal distribution, and the Friedman test will be used for measurements not showing normal distribution. In order to determine which groups the difference originates from, the t-test will be used for dependent groups in measurements showing normal distribution, and the Wilcoxon Sequential Signs test will be used for measurements not showing normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* No communication problems,
* Individuals diagnosed with cancer

Exclusion Criteria:

* Getting worse or dying during the research process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain levels of cancer patients will be evaluated using VAS. | 2 months
  Pain levels of cancer patients
Anxiety levels of cancer patients will be evaluated using the "State Anxiety Scale". | 2 months
  Anxiety levels of cancer patients
Psychological resilience levels of cancer patients will be evaluated using the "Brief Psychological Resilience Scale". | 2 months
  Psychological resilience levels of cancer patients

IPD SHARING:
Plan to Share IPD: No